CLINICAL TRIAL: NCT00732745
Title: Phase I/II Study of the Combination of Oxaliplatin / Docetaxel and ZACTIMA for the Treatment of Advanced Cancers of the Esophagus and Gastroesophageal Junction
Brief Title: Vandetanib, Oxaliplatin, and Docetaxel in Advanced Cancer of the Esophagus or Gastroesophageal Junction
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lost funding for Phase II portion of study
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE6507; P30CA043703 (NIH); CASE-6507 (Other: Case Comprehensive Cancer Center); NCT01019304 (obsolete NCT alias)
Record Dates: First submitted 2008-08-09; First posted 2008-08-12 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; adenocarcinoma of the gastroesophageal junction; squamous cell carcinoma of the esophagus; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Docetaxel; Oxaliplatin; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase II arm I (Experimental): Patients receive docetaxel IV over 1 hour on days 1 and 8, oxaliplatin IV over 2 hours on day 1, and oral vandetanib (at the maximum tolerated dose determined in phase I) once daily on days 1-21. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease may continue to receive vandetanib beyond 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: oxaliplatin; Drug: vandetanib
- Phase II arm II (Active Comparator): Patients receive docetaxel and oxaliplatin as in arm I. Patients also receive an oral placebo once daily on days 1-21. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease may continue to receive vandetanib beyond 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: oxaliplatin; Other: placebo

INTERVENTIONS:
Drug: docetaxel — Given IV
Drug: oxaliplatin — Given IV
Drug: vandetanib — Given orally
  Arms: Phase II arm I
Other: placebo — Given orally
  Arms: Phase II arm II

SUMMARY:
RATIONALE: Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as oxaliplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether vandetanib is more effective than a placebo when given together with oxaliplatin and docetaxel in treating advanced cancer of the esophagus or gastroesophageal junction.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of vandetanib when given together with oxaliplatin and docetaxel and to see how well it works in treating patients with advanced cancer of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of vandetanib when administered with oxaliplatin and docetaxel in patients with advanced cancer of the esophagus or gastroesophageal junction. (Phase I)
* To evaluate the toxicity of this regimen in these patients. (Phase I)
* To determine the progression-free survival of these patients. (Phase II)

Secondary

* To determine the response rate in patients treated with oxaliplatin and docetaxel with or without vandetanib. (Phase II)
* To determine the overall survival of patients treated with these regimens. (Phase II)
* To determine the toxicity of these regimens in these patients. (Phase II)
* To determine whether tumor characteristics (e.g., EGFR/ErbB2 expression, activation and mutational status of the EGFR and ErbB2 pathway [total and phosphorylated EGFR and ErbB2, mutational and FISH analysis] and tumoral expression of HIF1-alpha) may have an association with response and outcome. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of vandetanib followed by a randomized phase II study.

Patients are stratified according to histology (adenosarcoma vs squamous cell carcinoma) and prior neoadjuvant/adjuvant chemotherapy/chemoradiotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms. Patients in phase I receive treatment as in phase II arm I.

* Phase II arm I: Patients receive docetaxel IV over 1 hour on days 1 and 8, oxaliplatin IV over 2 hours on day 1, and oral vandetanib (at the maximum tolerated dose determined in phase I) once daily on days 1-21. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease may continue to receive vandetanib beyond 8 courses in the absence of disease progression or unacceptable toxicity.
* Phase II arm II: Patients receive docetaxel and oxaliplatin as in arm I. Patients also receive an oral placebo once daily on days 1-21. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease may continue to receive vandetanib beyond 8 courses in the absence of disease progression or unacceptable toxicity.

Patients enrolled in phase II submit baseline tumor tissue samples for correlative laboratory studies, including analysis of EGFR and ErbB2 by mutational, FISH, and IHC analysis and HIF1-alpha expression by IHC analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced adenocarcinoma or squamous cell carcinoma of the esophagus or gastroesophageal junction

  * Patients with locally advanced, unresectable disease are eligible provided they failed prior radiation-based therapy
* At least one measurable lesion
* No active CNS metastases as indicated by clinical symptoms, cerebral edema, or progressive growth

  * Patients with a clinical history of CNS metastases or cord compression are eligible provided they have been definitively treated and are clinically stable for ≥ 4 weeks (if treated with whole brain irradiation) or for ≥ 2 weeks (if treated with gamma knife therapy)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 12 weeks
* Hemoglobin > 9.5 g/dL
* ANC > 1,500/μL
* Platelets > 100,000/μL
* Total bilirubin normal
* Creatinine < 1.5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 30 mL/min
* AST, ALT, and alkaline phosphatase (AP) must meet one of the following criteria:

  * AST or ALT ≤ 5 times ULN AND AP normal
  * AST or ALT ≤ 1.5 times ULN AND AP ≤ 2.5 times ULN
  * AST or ALT normal AND AP ≤ 5 times ULN
* Potassium between 4 mmol/L and the upper limit of CTCAE grade 1 (supplementation allowed)
* Calcium (ionized or adjusted for albumin) and magnesium normal (supplementation allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No significant cardiovascular events within the past 3 months, including the following:

  * Myocardial infarction
  * Superior vena cava syndrome
  * NYHA class II-IV congestive heart failure
* No cardiac disease that, in the opinion of the investigator, may increase the risk of ventricular arrhythmia
* No prior arrhythmia (e.g., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (CTCAE grade 3)

  * Atrial fibrillation allowed provided it is controlled with medication
* No asymptomatic sustained ventricular tachycardia
* No hypertension not controlled by medical therapy (i.e., systolic blood pressure [BP] > 160 mm Hg or diastolic BP > 100 mm Hg)
* No QTc prolongation with other medication that required discontinuation of that medication
* No congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age
* QTc is < 480 with Bazett's correction on screening ECG at baseline
* No presence of left bundle branch block
* No active diarrhea > CTC grade 1
* No prior severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No prior allergic reactions to compounds of similar chemical or biologic composition to study drugs
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, would preclude study participation
* No other malignancy within the past 5 years, except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current PSA of < 1.0 mg/dL on 2 successive evaluations ≥ 3 months apart, with the most recent evaluation performed within the past 4 weeks
* No peripheral neuropathy > grade 1
* No blood donation during and for 3 months after completion of study treatment
* No severe or uncontrolled systemic disease or other medical condition, including mental illness or substance abuse, that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No prior systemic therapy for metastatic disease

  * Prior chemotherapy given as part of a definitive treatment plan (e.g., neoadjuvant or adjuvant chemotherapy or concurrent chemoradiotherapy) allowed
* More than 6 months since prior oxaliplatin and docetaxel as neoadjuvant or adjuvant therapy
* More than 4 weeks since prior major surgery, chemotherapy, radiotherapy, investigational agents, or other cancer therapy
* No prior anti-VEGF or EGFR therapy, including bevacizumab
* More than 2 weeks since prior and no concurrent potent CYP3A4 inducers (e.g.,rifampin, rifabutin, phenytoin, carbamazepine, phenobarbital, and Hypericum perforatum [St. John's wort])
* More than 2 weeks since prior and no concurrent medications known to cause QTc prolongation or to induce torsades de pointes
* No other concurrent chemotherapy, systemic antineoplastic therapy, or investigational therapy
* No concurrent radiotherapy, unless for local control of bone pain
* No concurrent cold cap or iced mouth rinses for prevention of alopecia or stomatitis
* No concurrent routine prophylactic use of granulocyte colony-stimulating factor (G-CSF) or pegfilgrastim
* No concurrent vitamin B6 supplementation, except as part of a standard multivitamin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vandetanib when administered with oxaliplatin and docetaxel (Phase I) | Each cycle of treatment consists of 21 days. Dose-limiting toxicities will be defined during cycle 1 of therapy. Patients will need to be observed for at least 2 cycles. A maximum of eight cycles of chemotherapy will be allowed.
Progression-free survival (Phase II) at 5 months | at 5 months

SECONDARY OUTCOMES:
Response rate (Phase II) | Tumor assessment will be performed after even treatment cycles every 6 weeks.
Overall survival (Phase II) | follow for life
Toxicity of oxaliplatin and docetaxel in combination with vandetanib or placebo (Phase II) | Day 8 and 15 of each treatment cycle and follow up (every 8 weeks) after chemotherapy.
Correlation of tumor characteristics and tumoral expression with response and outcome (Phase II) | Tumor assessment will be performed after even treatment cycles every 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Halmos B, Jia Y, Bokar JA, Fu P, Adelstein DJ, Juergens R, Rodal MB, Dowlati A. A Phase I study of the combination of oxaliplatin/docetaxel and vandetanib for the treatment of advanced gastroesophageal cancer. Invest New Drugs. 2013 Oct;31(5):1244-50. doi: 10.1007/s10637-013-9945-8. Epub 2013 Apr 4. PMID 23553066